CLINICAL TRIAL: NCT07101770
Title: Development and Validation of a Prediction Model for Adverse Pregnancy Outcomes in Women With Aplastic Anemia
Brief Title: A Prediction Model in Pregnant Women With Aplastic Anemia
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Lanzhou University Second Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); General Hospital of Ningxia Medical University (Other); Peking Union Medical College Hospital (Other); Peking University Third Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Wuhan TongJi Hospital (Other); Peking University First Hospital (Other); Chinese PLA General Hospital (Other); Second Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Soochow University (Other); Qilu Hospital of Shandong University (Other); Shanxi Provincial People's Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Shandong Provincial Hospital (Other Government); Shanxi Bethune Hospital (Other); Yantai Yuhuangding Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Principal Investigator, Peking University People's Hospital
Other Study IDs: 2025PHB251-001
Record Dates: First submitted 2025-07-02; First posted 2025-08-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Aplastic Anemia; Pregnancy; Prediction Model
Keywords: aplastic anemia; pregnancy; prediction model
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with adverse pregnancy outcomes
  Interventions: Other: A combined retrospective and prospective observational follow-up
- without adverse pregnancy outcomes
  Interventions: Other: A combined retrospective and prospective observational follow-up

INTERVENTIONS:
Other: A combined retrospective and prospective observational follow-up — A combined retrospective and prospective observational follow-up

SUMMARY:
Aplastic anemia (AA) is a rare haematologic disorder characterized by bone marrow failure and pancytopenia. Its occurrence during pregnancy is exceedingly rare but poses significant risks, including maternal hemorrhage, infections, and perinatal complications such as preterm birth and fetal growth restriction. Consequently, pregnancy with AA is highly perilous for both mothers and infants. Early management is critical to ensure the health of both the mother and the baby. However, there are currently no predictive tools available to assess adverse outcomes in pregnant women with AA. Our center plans to conduct a multicenter, combined retrospective and prospective cohort study.

DETAILED DESCRIPTION:
The gestational period, a physiological condition linked to elevated physiological stress, induces significant cardiac remodeling and systemic hemodynamic adaptations in maternal organisms. AA, a rare but life-threatening hematologic disorder characterized by pancytopenia and bone marrow hypoplasia, poses profound challenges during pregnancy, with significant risks of maternal and perinatal morbidity and mortality. Physiological adaptations in pregnancy, including hemodilution and increased metabolic demands, exacerbate AA-related hematologic deficits, elevating risks of severe anemia, thrombocytopenia-related hemorrhage, and immunosuppression-associated infections. These outcomes underscore the critical need for dynamic risk stratification and tailored interventions.

Currently, most cohort studies on pregnant women with AA in China are retrospective, single-center studies with small sample sizes, resulting in insufficient data and a lack of multicenter, prospective cohort studies.

This study is a multicenter, retrospective and prospective observational study that will enroll pregnant women with aplastic anemia. It will collect baseline patient information and diagnostic data, conduct regular prospective follow-ups via questionnaires, telephone interviews, video consultations, online platforms, and in-person visits, and record treatment regimens, comorbidities, and prognostic outcomes. The study aims to provide comprehensive data on the epidemiology and clinical outcomes of pregnant women with aplastic anemia in China, and aimed to develop and validate a predictive model for adverse pregnancy outcomes in pregnant women with AA, with the goal of guiding early clinical decision-making and improving their overall health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women who had aplastic anemia before pregnancy
2. pregnant women with newly diagnosed aplastic anemia during pregnancy

Exclusion Criteria:

1. age less than 20 years
2. without coagulation series results
3. termination of pregnancy before 20 weeks of gestation
4. multiple pregnancy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population included pregnant women with aplastic anemia 20 years of age or older. This study was conducted in strict accordance with the Declaration of Helsinki and was approved by ethics committees or central institutional review boards of the Peking University People's Hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-27 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse pregnancy outcomes | From the first visit to hospital during pregnancy to 42 days after delivery
  Incident of adverse pregnany outcomes include at least one of the conditions as follows:
  placental abruption (ultrasound to detect a retroplacental hematoma), amniotic fluid embolism (elevated fetal squamous cells, vernix, or meconium in maternal blood; prolonged PT, APTT, low fibrinogen, and elevated D-dimers), postpartum hemorrhage (≥500 mL blood loss within 24 hours of vaginal delivery or ≥1000 mL after cesarean delivery), postpartum infection (fever, leukocytosis, etc), maternal mortality, stillbirths (fetal death occurring at ≥20 weeks of gestation), preterm birth (delivery at <37 weeks of gestation), low birthweight ( a newborn with birth weight <2500 g), fetal growth restriction (a fetus with estimated fetal weight or abdominal circumference <10th percentile for gestational age), neonatal intensive care unit admission, or neonatal mortality (death of a live-born infant within the first 28 days of life).

SECONDARY OUTCOMES:
Neonatal Apgar Score | within 10 minutes after birth
  Apgar 1-minute, 5-minute, 10-minute scores

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided